CLINICAL TRIAL: NCT06634680
Title: Effects of Different Parental Involvement on Anxiety and Delirium in Children Undergoing Elective ENT Surgery
Brief Title: Effects of Different Parental Involvement on Anxiety and Delirium
Status: Completed | Type: Observational
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 04- 2024/15
Record Dates: First submitted 2024-10-02; First posted 2024-10-10 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-10

CONDITIONS: Anxiety State; Child Behavior
Keywords: anxiety; children; anesthesia,general
MeSH Terms: conditions — Anxiety Disorders; Child Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group Child Preference: The children will prefer parents (mother or father) who will accompany them in the preoperative holding area and at induction.
  Interventions: Procedure: Procedure: Selection of parent(mother or father) according to children preference
- Group Both Parents: Both parents will accompany the child in the preoperative holding area and at induction.
  Interventions: Procedure: Procedure: Both parents will accompany the children.

INTERVENTIONS:
Procedure: Procedure: Selection of parent(mother or father) according to children preference — Children will choose the parent who will accompany them.
  Groups: Group Child Preference
Procedure: Procedure: Both parents will accompany the children. — Both parents will accompany the children.
  Groups: Group Both Parents

SUMMARY:
Induction of anesthesia in surgical procedures can be a distressing process for both children and their parents. Nonpharmacological behavioral interventions, unlike sedative medications, can reduce children's anxiety without adverse effects. The effect of having both parents present during anesthesia induction on children's anxiety and parents' anxiety has not yet been documented.

This study will aim to evaluate the effect of having both parents present during anesthesia induction on children's and parental anxiety during the perioperative period.

DETAILED DESCRIPTION:
Surgery can be very stressful for patients, especially children. Studies show that 50-75% of children experience fear and anxiety when undergoing surgery and being put under anesthesia. This anxiety can have adverse effects on their recovery, leading to more extended hospital stays, increased pain, and behavioral issues. To address this, various medical and non-medical approaches are used to ease children's fears. One such approach is allowing parents to be with their children until the anesthesia takes effect. This study aims to assess how having both parents present during this time impacts the child's anxiety levels.

The effect of parental presence on the anxiety of children and parents was studied in various studies. Whether both parents affect anxiety has not been studied yet. In this study the investigators will evaluate the anxiety of children by using mYPAS.

ELIGIBILITY:
Inclusion Criteria:

* 80 children of both sex, aged 5-12 years with ASA physical Status I-II will be enrolled

Exclusion Criteria:

* Mentally challenged
* Deaf Child
* Cerebral Palsy
* Premedicated Child
* Language Problem
* Uncooperative
* History of psychiatric disease in children or the parents
* Previous surgery or anesthesia history

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study included 80 children of both genders, aged 5-12 years, who underwent day-case surgery in the otorhinolaryngology clinic
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Patients anxiety-Modified Yale Preoperative Anxiety Scale (mYPAS) of the children undergoing elective surgery under general anesthesia. | Perioperative period
  The mYPAS will be used to evaluate the anxiety level of children. The mYPAS is an observational measure of preoperative anxiety consisting of 27 items in 5 domains (activity, emotional expressivity, state of arousal, vocalization, and use of parents). The adjusted mYPAS total score ranges from 23.3 to 100, with higher scores indicating greater anxiety.

SECONDARY OUTCOMES:
Emergence delirium-Pediatric Anesthesia Emergence Delirium Scale (PAEDS) | Perioperative period
  Pediatric Anaesthesia Emergence Delirium (PAED) scale consists of 5 criteria (eye contact, purposeful movement, awareness of environment, restlessness, inconsolability) that are scored using a 5-point scale. The scores of each criterion are added to make a total score. The score changes 0-20. Scores above 10 indicate delirium, while scores below 10 indicate no delirium.
Parent anxiety-STAI | Perioperative period
  The State-Trait Anxiety Inventory (STAI) was used to evaluate the anxiety level of the parents. The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety. It has 20 items for assessing trait anxiety and 20 for state anxiety. State anxiety items include: "I am tense; I am worried" and "I feel calm; I feel secure." Trait anxiety items include: "I worry too much over something that really doesn't matter" and "I am content; I am a steady person." All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Rafet YARIMOGLU, Principal Investigator — Karaman Training and Research Hospital
Locations (1):
- Rafet YARIMOGLU, Karaman, Karaman, Turkey (Türkiye)

REFERENCES:
- [Derived] Yarimoglu R, Sezgin A, Duran A, Yucedag F, Basaran B. The Impact of the Presence of Both Parents on Perioperative Anxiety in Children Undergoing Adenotonsillectomy Surgery: A Randomized Clinical Trial. Acta Anaesthesiol Scand. 2026 Jan;70(1):e70167. doi: 10.1111/aas.70167. PMID 41423202